CLINICAL TRIAL: NCT05211427
Title: Expression of Bitter Taste Receptors in Oropharynx Carcinoma
Brief Title: Bitter Taste Receptors in Oropharynx Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Hummel (Other)
Responsible Party: Sponsor-Investigator, Thomas Hummel, Director, Interdisciplinary Smell and Taste Centre, Technische Universität Dresden
Organization: Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ENTASTE
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patients with oropharynx cancer
  Interventions: Procedure: Biopsy
- Healthy subjects (Experimental): Patients with non malignant pharynx pathology
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsy of an oropharynx tumor or of a healthy oropharynx mucosa

SUMMARY:
The aim of this work is to investigate the expression of the bitter taste receptors in p16-positive and negative oropharyngeal carcinomas (in comparison to healthy, local tissue).

DETAILED DESCRIPTION:
Goal setting The aim of this work is to investigate the expression of the bitter taste receptors in p16-positive and negative oropharyngeal carcinomas (in comparison to healthy, local tissue).

The hypothesis is that oropharyngeal carcinomas express TAS2Rs and that their stimulation can induce apoptosis. The lower expression of certain TAS2Rs in the tumor cells could represent protection from apoptosis by stimulation with the bitter ligands. Alternatively, it could polymorphisms of the bitter taste receptors, which can influence their function independently of the expression. In order to address the question of general bitter sensitivity in more detail, the investigators are planning to carry out a bitter taste test on the test subjects.

methodology As this is a pilot study, the investigators limit the number of subjects to 10 patients with p-16 positive and negative oropharyngeal squamous cell carcinoma and 10 patients with acute recurrent tonsillitis or other benign pathology in pharynx. The expression analysis is carried out using qPCR and possibly immunohistochemical methods. Taste strips are used for the taste tests.

Cognitive interest The results of this study will provide important insight into the pathophysiology of oropharyngeal cancers and possibly all TAS2R-expressing cancers. In addition, this and further studies can create a theoretical basis for new therapeutic methods for this group of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Oropharynx SCC for the patient group
* signed informed consent for all

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Expression of TAS2-Receptors | The day of surgery and the day before
  relative concentration of TAS2Rs in mucosa and tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Smell and Taste Center, University Klinik Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the regulations of the publishing journal